CLINICAL TRIAL: NCT06015854
Title: A Phase II Study to Determine the Efficacy and Safety of Vvax001, a Therapeutic Semliki Forest Virus Based Cancer Vaccine, in Patients With HPV-16 Induced Grade 3 Cervical Intraepithelial Neoplasia
Brief Title: Vvax001 Cancer Vaccine in Premalignant Cervical Lesions - Phase II
Acronym: Vvax
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other); ViciniVax B.V (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vvax001-UMCG-02
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: CIN3; Cervical Intraepithelial Neoplasia; Cervical Intraepithelial Neoplasia Grade 3; HPV 16 Infection
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV16+ CIN3 (Experimental): Patients with histological proven HPV16-positive cervical intraepithelial neoplasia grade 3.
  Interventions: Biological: Vvax001 therapeutic cancer vaccine

INTERVENTIONS:
Biological: Vvax001 therapeutic cancer vaccine — Patients will receive three immunizations, with an interval of 3 weeks between each immunization at weeks 0, 3 and 6. Each vaccination will be given as two injections; 1 injection in each leg. The injections will be administered intramuscularly in the upper legs, preferably in the m. vastus lateralis.

SUMMARY:
This is an open label phase II study in patients with newly diagnosed human papilloma virus type 16 (HPV16) induced cervical intraepithelial neoplasia grade 3 (CIN3). Patients will be treated with three doses of Vvax001 immunization with an interval of 3 weeks between each immunization to induce histopathological regression and HPV clearance. Regression of CIN3 lesions will be monitored using colposcopy in week 9, week 17 and week 25. When complete regression of the CIN3 lesion is observed by colposcopy, a biopsy will be taken in week 25 to confirm regression histologically. A positive histologic regression is defined as a reduction from CIN3 to CIN1 or no dysplasia. Patients with a complete regression will not undergo the standard-of-care loop excision of the transformation zone (LETZ) and will be followed-up after the study by cytology at 3, 6 and 12 months. If complete regression has not occurred by 25 weeks, a standard-of-care LETZ will be performed.

DETAILED DESCRIPTION:
Human papillomavirus (HPV) infection is the most important cause of premalignant cervical disease. Current treatment for premalignant HPV-induced genital lesions primarily relies on surgery, which can be discomforting and carries a risk of complications like bleeding, cervical stenosis and/or incompetence which may lead to infertility and partus prematuris/immaturis. Above all, it does not necessarily eradicate the underlying HPV infection completely.

Therapeutic immunization is a very attractive alternative to the current treatment options for precancerous lesions and (invasive) cancer. The immune cells induced by cancer immunotherapy can target the tumor cells and kill them. When long-lasting immunity is induced the immunotherapy may prevent recurrence of the disease. Therefore, the approach taken in this study is to immunize with a replication-incompetent Semliki Forest Virus (SFV) vector encoding HPV-derived tumor antigens. Intramuscular immunization with these replication-incompetent SFV particles (Vvax001) is aimed at eliciting a therapeutic anti-tumor response.

A phase I study has been conducted in which vaccination with Vvax001 induced HPV16-E6,7-specific immune responses in women previously treated for cervical intraepithelial neoplasia (CIN) or cervical cancer (CC). Intramuscular immunization with Vvax001 was well tolerated, showing only mild to moderate local adverse reactions. Altogether, the data of this study justify testing of Vvax001 in CIN3 patients in the current phase II study.

In this open label phase II study patients with newly diagnosed HPV16 induced cervical intraepithelial neoplasia grade 3 (CIN3) will receive three bilateral intramuscular immunizations of Vvax001 (5x107 infectious particles [IP]) with an interval of 3 weeks between vaccinations at week 0, week 3 and week 6.

Patients will be monitored for regression of CIN3 lesions by colposcopy and digital imaging at week 9, week 17 and week 25. When complete regression of the CIN3 lesion is observed by colposcopy, a biopsy will be taken in week 25 to confirm regression and no LETZ will be performed. If complete regression has not occurred by 25 weeks, the standard-of-care LETZ will be performed. If progression of the CIN3 lesion is observed during the 25 week interval, a biopsy will be taken to confirm pathological progression. If pathological progression has occurred, patients will immediately undergo a LETZ. If no pathological progression has occurred, patients will continue to be monitored by colposcopy.

Patients with a complete regression will be followed-up by cytology at 3, 6 and 12 months after exit from the study. Hereafter, patients will be monitored through regular screening programs.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed HPV16-positive CIN3.
* Age of 18 years and older.
* Patients of child-bearing potential should test negative using a serum pregnancy test and agree to utilize effective contraception during the entire treatment and follow-up period of the study.
* Written informed consent according to local guidelines.

Exclusion Criteria:

* PAP5 lesions.
* Previously undergone treatment for CIN lesions.
* Adenocarcinoma in situ within CIN3 lesion.
* History of an autoimmune disease or other systemic intercurrent disease that might affect the immunocompetence of the patient, or current or prior use (4 weeks before start of the study) of high dose immunosuppressive therapy.
* History of a malignancy except curatively treated low-stage tumors with a histology that can be differentiated from the cervical cancer type.
* Participation in a study with another investigational drug within 30 days prior to the enrolment in this study.
* Clinically significant findings as judged by the Investigator on screening/study entry including those from the Biochemistry, Hematology and urinalysis performed at baseline.
* Any condition that in the opinion of the investigator could interfere with the conduct of the study.
* Pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2024-02-06 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy of Vvax001 | At week 25 (19 weeks after the last immunization)
  Clinical efficacy is determined by a pathological regression of the premalignant CIN3 lesion in pre- versus post-treatment tissue samples. A positive histologic regression is defined as a reduction from CIN3 to CIN1, or a reduction from CIN3 to no dysplasia.

SECONDARY OUTCOMES:
Immunogenicity of Vvax001 | At weeks 7, 9, 17 and 25, respectively 1 week, 3 weeks, 11 weeks and 19 weeks after the last vaccination
  HPV-16 E6,7-specific T-cell immune responses in the peripheral blood will be measured by IFN-y ELISPOT
HPV 16 clearance | Week 25 (19 weeks after the last immunization)
  Standard HPV testing by molecular analysis will be performed on tissue collected during the last study visit.
Side effects/ adverse events | up to 19 weeks after the last immunization
  To monitor the side effects/ adverse events related to intramuscular administration of Vvax001. Toxicity will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen (UMCG), Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided